CLINICAL TRIAL: NCT02557893
Title: Effects of Exercise on Back Pain in Pregnancy
Brief Title: Effects of Resistance Exercise During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01NR008131 (NIH)
Record Dates: First submitted 2015-09-09; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy
MeSH Terms: interventions — Resistance Training; Educational Status; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resistance exercise (Experimental): Resistance exercise involved 12 weeks of weight lifting exercise
  Interventions: Behavioral: Resistance exercise
- Wait list (Sham Comparator): Wait list participants were tested on the outcomes during their pregnancy and were eligible to participate in a post-partum supervised exercise program. The wait list participants formed a no treatment control group.
  Interventions: Other: Wait list
- Pregnancy education (Placebo Comparator): Maternity nurses taught six bimonthly pregnancy education classes (~20 per class) which covered several topics including information about what to expect during normal labor and delivery, common interventions during delivery (medications, induction, Cesarean delivery), parenting skills needed for baby care, breastfeeding, baby and child cardiopulmonary resuscitation, typical child development and communicating with infants. No physical activity education was included in the curriculum. The pregnancy education participants formed an attention control group.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Resistance exercise — Resistance exercise involved 12-weeks of strength training twice per week
  Arms: Resistance exercise
Other: Education — Bimonthly pregnancy education classes
  Arms: Pregnancy education
Other: Wait list — Wait list participants were tested on the outcomes during their pregnancy and were eligible to participate in a post-partum supervised exercise program. The wait list participants formed a no treatment control group.
  Arms: Wait list

SUMMARY:
Pregnant women at increased risk for back pain were studied during the second trimester and randomized to12-weeks of resistance exercise, education or waitlist. Several outcomes were assessed including physical function, quality of life and mood.

DETAILED DESCRIPTION:
A parallel group trial was completed at a single site. Second trimester women (n=134) were randomly assigned (in blocks of 3) to 12-weeks of wait list, bi-monthly pregnancy education classes or twice weekly low-to-moderate intensity resistance training. Resistance training involved one abdominal exercise with no external load and five exercises with an external load that gradually progressed (leg extension, leg press, arm lat pull, leg curl, and lumbar extension). Several outcomes were assessed including physical function, quality of life and mood.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and able to complete baseline testing during gestational week 21 to 25 of pregnancy.

Exclusion Criteria:

* Regular resistance exercise training (≥ twice per week during the past month)
* an orthopedic or cardiovascular limitation
* a psychiatric disorder
* or had in the current or a prior pregnancy any of the following:

  * two or more miscarriages
  * premature labor
  * placental previa,
  * poor fetal growth,
  * low pre-pregnancy body weight (BMI < 17.5)
  * a multiple birth pregnancy
  * pre-eclampsia
  * preterm rupture of membranes
  * uterine growth retardation
  * incompetent cervix/cerclage
  * recurrent vaginal bleeding
  * anemia or
  * diabetes.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Physical function measured with physical tests such as time to make a bed, get up and down off the floor and pick up scarves from the floor. | Change from week 21 to 35 of pregnancy
  The intervention occurred from weeks 22 to 34 of pregnancy and the outcomes were measured the week before and after the intervention.
Quality of life measured using the Short Form 36 Healthy Survey. | Change from week 21 to 35 of pregnancy
  The intervention occurred from weeks 22 to 34 of pregnancy and the outcomes were measured the week before and after the intervention.
Mood measured using the Profile of Mood States questionnaire. | Change from week 21 to 35 of pregnancy
  The intervention occurred from weeks 22 to 34 of pregnancy and the outcomes were measured the week before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O'Connor, Ph.D., Principal Investigator — University of Georgia

REFERENCES:
- [Result] O'Connor PJ, Poudevigne MS, Cress ME, Motl RW, Clapp JF 3rd. Safety and efficacy of supervised strength training adopted in pregnancy. J Phys Act Health. 2011 Mar;8(3):309-20. doi: 10.1123/jpah.8.3.309. PMID 21487130
- [Derived] O'Connor PJ, Poudevigne MS, Johnson KE, Brito de Araujo J, Ward-Ritacco CL. Effects of Resistance Training on Fatigue-Related Domains of Quality of Life and Mood During Pregnancy: A Randomized Trial in Pregnant Women With Increased Risk of Back Pain. Psychosom Med. 2018 Apr;80(3):327-332. doi: 10.1097/PSY.0000000000000559. PMID 29394188